CLINICAL TRIAL: NCT02940002
Title: A 28-day, Double-blind, Randomized, Reference-controlled Psoriasis Plaque Test to Evaluate the Efficacy and Safety of Two Different BAY1003803 Formulation Types in 2 Concentrations Each in Treatment of Symptomatic Volunteers With Plaque-type Psoriasis
Brief Title: BAY1003803 Formulation Comparison in Open Psoriasis Plaque Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17012; 2016-000962-47 (EudraCT Number)
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
Keywords: Plaque form psoriasis vulgaris
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- BAY1003803 0.1% lipophilic cream (Experimental): BAY1003803 0.1% lipophilic cream (on plaque and healthy skin)
  Interventions: Drug: BAY1003803
- BAY1003803 0.1% ointment (Experimental): BAY1003803 0.1% ointment (on plaque and healthy skin)
  Interventions: Drug: BAY1003803
- BAY1003803 0.01% lipophilic cream (Experimental): BAY1003803 0.01% lipophilic cream (on plaque and healthy skin)
  Interventions: Drug: BAY1003803
- BAY1003803 0.01% ointment (Experimental): BAY1003803 0.01% ointment (on plaque and healthy skin)
  Interventions: Drug: BAY1003803
- Clobetasol propionate (Active Comparator): Clobetasol propionate ointment 0.05 % (on plaque and healthy skin)
  Interventions: Drug: Clobetasol propionate
- Betamethasone/calcipotriene (Active Comparator): Betamethasone/calcipotriene ointment 0.05 %/0.005% (on healthy skin)
  Interventions: Drug: Betamethasone/calcipotriene

INTERVENTIONS:
Drug: BAY1003803 — Simultaneous application of 10μl on psoriasis plaque and on healthy skin for 4 weeks and evaluation of pharmacodynamic effect
  Arms: BAY1003803 0.01% lipophilic cream; BAY1003803 0.01% ointment; BAY1003803 0.1% lipophilic cream; BAY1003803 0.1% ointment
Drug: Clobetasol propionate — Simultaneous application of 10μl on psoriasis plaque and on healthy skin for 4 weeks and evaluation of pharmacodynamic effect
  Arms: Clobetasol propionate
Drug: Betamethasone/calcipotriene — Simultaneous application of 10μl on healthy skin for 4 weeks and evaluation of pharmacodynamic effect
  Arms: Betamethasone/calcipotriene

SUMMARY:
To explore the efficacy and safety of four BAY1003803 formulations by means of a within subject comparison in an open Psoriasis Plaque Test

ELIGIBILITY:
Inclusion Criteria:

* Male and female (non-childbearing potential) volunteer with stable plaque-type psoriasis, but otherwise healthy
* Age: 18-64 years

Exclusion Criteria:

* Severe disease within the last 4 weeks prior to the first study drug administration as determined by the investigator
* Any topical antipsoriatics on plaques potentially to be treated in this trial (including corticosteroids, vitamin D analogues, immunomodulators, retinoids, dithranol and tar, except for salicylic acid (Pretreatment) in the 4 weeks before first treatment and/or planned during the trial, except for allowed topical treatment on the face, ears and scalp
* Systemic treatment depending on kind of treatment within 4 weeks and 6 months prior and/or planned during the trial
* Treatment with concomitant medication that may affect and provoke or aggravate psoriasis, e.g. antimalarial drugs, lithium, beta-blockers or angiotensin-converting-enzyme inhibitors (AEC inhibitors) unless on a stable dose for 3 months before study medication initiation
* Clinico-chemical parameters of clinically significant deviation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Change in infiltrate thickness from day 1 to day 29 measured by sonography using 22 MHz B mode ultrasound | Day 1 to 29

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Germany (3):
  - Hamburg, Hamburg
  - Schwerin, Mecklenburg-Vorpommern
  - Bochum, North Rhine-Westphalia